CLINICAL TRIAL: NCT03905382
Title: Exploring the Experiences and Views of Patients, Their Carers' and Health Care Providers on the Use of Modems in Managing Patients Receiving Domiciliary Non-invasive Ventilation (NIV): a Qualitative Study
Brief Title: Non-invasive Ventilator Modems: a Qualitative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Stephanie Mansell, Consultant Physiotherapist, Royal Free Hospital NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9816
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Ventilatory Failure
Keywords: Technology; Modems; Qualitative Research
MeSH Terms: conditions — Hypoventilation | interventions — Evaluation Studies as Topic

STUDY DESIGN:
Intervention Model Description: Single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Qualitaitve (Other): Qualitaitve
  Interventions: Other: Qualitative

INTERVENTIONS:
Other: Qualitative — Focus group and 1:1 telephone interviews

SUMMARY:
Advances in technology has meant that domiciliary non-invasive (NIV) devices can be remotely monitored via modems in patients' homes. Possible benefits and challenges of modem technology have yet to be established. This study explored the perspectives and experiences of patients, their carers' and health care professionals (HCPs) on the addition of modem technology in managing home NIV patients.

DETAILED DESCRIPTION:
The aim of this study is to consider the opinions of patients, their carers' and health care providers on the addition of using modem technology in the management of patients with hypercapnic respiratory failure receiving domiciliary NIV.

Objectives

1. To investigate the experience of patients receiving domiciliary NIV with modem technology and how this compares to NIV treatment without a modem
2. To investigate the experience of carers' of patients receiving domiciliary NIV with modem technology and how this compares to NIV treatment without a modem
3. To gain opinions of health care providers on the use of modem technology in caring for patient with ventilatory failure and how this compares to delivering home NIV treatment without a modem 4.2 Outcome The outcome of this study will inform future service development of home NIV services to ensure they are designed with service users' preferences in mind.

ELIGIBILITY:
Inclusion Criteria:

Patients and carers •Patients and their carers who received treatment from the Royal Free London (RFL) domiciliary NIV service both pre and post modem installation will be eligible to be included in the study.

HCPs

•Staff who have experience of looking after patients with NIV both with and without modems will be able to take part in the study. Staff recruited will be currently working at RFL. We have been using modems for all of our patients with NIV since December 2014. Therefore rotational staff (e.g. registrars) working RFL will only have experience of looking after patients with modems on their NIV. To allow for this factor staff will be allowed to join the study even if their experience of looking after patients with NIV without modems is at other hospitals.

Exclusion Criteria:

* Patients under the care of the RFL domiciliary NIV service who have only had experience of treatment with a modem in situ will be excluded from the study.
* Patients who are unable to verbally communicate
* Patients who cannot have an "everyday" level conversation in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Focus groups, 1:1 telephone interviews | 18 months
  Modified thematic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Mansell, Principal Investigator — Royal Free London NHS FoundationTrust
Locations (1):
- Royal Free London NHS foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analysed during the current study are not publicly available in order to maintain participant anonymity, but are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Mansell SK, Kilbride C, Wood MJ, Gowing F, Mandal S. Experiences and views of patients, carers and healthcare professionals on using modems in domiciliary non-invasive ventilation (NIV): a qualitative study. BMJ Open Respir Res. 2020 Mar;7(1):e000510. doi: 10.1136/bmjresp-2019-000510. PMID 32161065